CLINICAL TRIAL: NCT02034227
Title: An Open-Label, Phase 1/Phase 2 Study to Evaluate the Safety, Tolerability, and Antitumor Activity of the DNA Minor Groove Binding Agent SG2000 in the Treatment of Advanced Chronic Lymphocytic Leukemia and Acute Myeloid Leukemia
Brief Title: Safety, Tolerability Study of SG2000 in the Treatment of Advanced Chronic Lymphocytic Leukemia and Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Spirogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL-2000-II-01
Record Dates: First submitted 2014-01-06; First posted 2014-01-13 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2015-11

CONDITIONS: Acute Myeloid Leukemia; Chronic Lymphocytic Leukemia
Keywords: leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia

ARMS (2):
- SG2000 - 15 µg/m2/day (Experimental): Cohort 1 - will commence at 15 µg/m2/day intravenous doses of SG2000 until Maximum Tolerated Dose is determined.
  Interventions: Drug: SG2000
- SG2000 - 30 µg/m2/day (Experimental): Cohort 2 - will commence at 30 µg/m2/day intravenous doses of SG2000 until Maximum Tolerated Dose is determined.
  Interventions: Drug: SG2000

INTERVENTIONS:
Drug: SG2000 — intravenous doses given on Days 1, 2, and 3 of each 21-day cycle (1 to 6 cycles).
  Other Names: DNA minor groove binding agent

SUMMARY:
The purpose of this study is to determine if the experimental drug, SG2000 is safe and tolerable in the treatment of participants with advanced chronic lymphocytic leukemia and acute myeloid leukemia whose standard treatment did not work, whose cancer came back or who are not candidates for other types of standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* male or female greater than or equal to 18 years of age
* have one of the following disease states: Acute Myeloid Leukemia (AML) (age <60 years) with relapsed/refractory disease; •Chronic Lymphocytic Leukemia (CLL) with relapsed disease following a fludarabine-based regimen or relapsed disease following an alkylator-based regimen
* are recovered from the acute adverse effects of prior therapies (excluding alopecia and Grade ≤2 neuropathy).
* have blast counts that can be controlled by the use of hydroxycarbamide (500 to 3000 mg daily).
* have adequate hepatic function and renal function
* have an estimated life expectancy of >3 months
* female subject must have a negative serum pregnancy result within 7 days before the start of the study; Both men and women must agree to use a medically acceptable form of contraception throughout the treatment period and for 3 months after discontinuation of treatment

Exclusion Criteria:

* are eligible for any standard therapy known to be life prolonging or life saving
* have diagnosis of AML French-American-British (FAB) classification (FAB) M3 (acute promyelocytic leukemia (APL))
* are receiving concurrent chemotherapy, radiotherapy, immunotherapy, biological or hormonal treatment for cancer.
* have undergone anticancer therapy including chemotherapy (except for hydroxycarbamide at a maximum daily dose of 3000 mg), endocrine therapy, immunotherapy, or the use of other investigational agents within 4 weeks before study entry.
* prior radiation therapy with volume of bone marrow treated over 25%.
* use of immunosuppressive therapy, including systemic steroids within 7 days before the first dose of SG2000.
* hyperleukocytosis (blast counts >30 000/mm3).
* history of allogeneic stem cell or solid organ transplantation.
* positive serology for human immunodeficiency virus (HIV), hepatitis B or hepatitis C or have HIV-AIDS, or active hepatitis B or C.
* history of other invasive malignancy within 3 years except for cervical carcinoma in situ, nonmelanomatous carcinoma of the skin or ductal carcinoma in situ of the breast that has been surgically cured.
* have any coexisting medical condition that will substantially increase the risk associated with the subject's participation in the study.
* have psychiatric disorders or altered mental status precluding understanding of the informed consent process and/or completion of necessary studies.
* have persistent Grade 2 or greater toxicities from any cause (except alopecia or peripheral neuropathy).
* are pregnant or breast-feeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2012-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of SG2000. | From 1st dose of SG2000 given on days 1, 2 and 3, every 21-days, for six 21-day cycles (approximately 16 weeks).
  The Maximum Tolerated Dose (MTD) will be determined based on the assessment of the dose-limiting toxicity (DLT) during the DLT period; period is defined as the time from the first dose intravenous doses of SG2000 for 3 consecutive days every 21 days for 1 to 6 cycles until unacceptable toxicity, consent withdrawal, or another reason to discontinue therapy intervenes.

SECONDARY OUTCOMES:
safety profile | day -1 to day- 21 for six 21-day cycles .
  Any subject who receives at least 1 dose of SG2000 will be evaluated for safety.
  Subjects will be monitored for adverse events (AEs) and will undergo safety assessments including full physical examination, vital sign assessment, Eastern Cooperative Oncology Group (ECOG) performance status assessment, and laboratory testing.
area under the concentration-time curve (AUC) | day-1 of each 21-day cycle (cycles 1 and 3) at the following time points: predose, 15 minutes (middle of infusion), 30 minutes(end of infusion), and at 10 minutes, 20 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, and 24 hours after the end of infusion.
  pharmacokinetic (PK) parameter, noncompartmental analysis will be performed to estimate the plasma pharmacokinetic (PK) parameters of SG2000. Area under the concentration-time curve (AUC).
Maximum plasma concentration (Cmax) | day-1 of each 21-day cycle (cycles 1 and 3) at the following time points: predose, 15 minutes (middle of infusion), 30 minutes (end of infusion), and at 10 minutes, 20 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, and 24 hours after the end of infusion.
  pharmacokinetic (PK) parameter -Cmax is the observed maximum plasma or serum concentration after administration
time to reach Cmax | day-1 of each 21-day cycle (cycles 1 and 3) at the following time points: predose, 15 minutes (middle of infusion), 30 minutes (end of infusion), and at 10 minutes, 20 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, and 24 hours after the end of infusion.
  pharmacokinetic (PK) parameter - time to reach Cmax.
terminal half life (T1/2), | day-1 of each 21-day cycle (cycles 1 and 3) at the following time points: predose, 15 minutes (middle of infusion), 30 minutes (end of infusion), and at 10 minutes, 20 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, and 24 hours after the end of infusion.
  pharmacokinetic parameter - terminal half life
hematology and serum chemistry | baseline, days 1,2,3,4,8,15, and 21 for six 21-day cycles.
  predictors of Vascular Leak Syndrome (VLS)
Physical examination | baseline, day-1 to day 21 for six 21-day cycles.
  predictors of Vascular Leak Syndrome (VLS)
Vital signs | baseline, day-1 to day-21 for six 21-day cycles.
  predictors of Vascular Leak Syndrome (VLS)
bone marrow aspirate | day-1 (predose), and day 8 of Cycles 1 and 3 , and day 1 of Cycles 2 and 4
pulse oximetry | baseline, day-1 to day-21 for six 21-day cycles.
  monitoring for Vascular Leak Syndrome (VLS)
electrocardiogram | days 1, 8, 15, 21, and at Day 22 after the last cycle or early termination.
bone marrow aspirate | day-1 (predose), and day- 8 of each 21-day cycle (cycles 1 and 3) and day -1 of cycles 2 and 4

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Duke University, Durham, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina